CLINICAL TRIAL: NCT01718158
Title: A Phase 3 Evaluation of Daclatasvir in Combination With Peginterferon Lambda-1a and Ribavirin (RBV) or Telaprevir in Combination With Peginterferon Alfa-2a and RBV in Patients With Chronic Hepatitis C Genotype 1b Who Are Treatment naïve or Prior Relapsers to Alfa/RBV Therapy (the STRUCTURE Study)
Brief Title: Efficacy and Safety Evaluation of a Regimen Consisting of Peginterferon Lambda-1a + Ribavirin + Daclatasvir (Lambda + RBV + DCV) in HCV Genotype 1b Treatment naïve Patients or Prior Relapsers to Peginterferon Alfa + Ribavirin (Alfa + RBV) Therapy
Acronym: STRUCTURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI452-021; 2011-005409-65 (EudraCT Number)
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon lambda-1a; peginterferon alfa-2a; Ribavirin; daclatasvir; telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peginterferon Lambda-1a + Ribavirin + Daclatasvir (Experimental): Peginterferon Lambda-1a 180 µg solution for subcutaneous injection, once a week for 24 Weeks
  Ribavirin 200 mg tablets [1000-1200 mg total daily dose: subjects should take either 400 mg (2 tablets for subjects < 75 kg) or 600 mg (3 tablets for subjects ≥ 75 kg) in the morning with food and 600 mg (3 tablets) in the evening with food] by mouth, twice daily, for 24 weeks
  Daclatasvir 60 mg tablets by mouth, once a day for 12 weeks
  Interventions: Biological: Peginterferon Lambda-1a; Drug: Ribavirin; Drug: Daclatasvir
- Peginterferon Alfa-2a + Ribavirin + Telaprevir (Experimental): Peginterferon Alfa-2a 180 µg solution for subcutaneous injection, once a week for 24 to 48 weeks depending on response
  Ribavirin 200 mg tablets [1000-1200 mg total daily dose: subjects should take either 400 mg (2 tablets for subjects < 75 kg) or 600 mg (3 tablets for subjects ≥ 75 kg) in the morning with food and 600 mg (3 tablets) in the evening with food] by mouth, twice daily, for 24 to 48 weeks depending on response
  Telaprevir 375 mg tablets [2250 mg total daily dose: subjects should take 750 mg (two 375 mg tablets) orally three times a day, approximately 7-9 hours apart) for 12 weeks
  Interventions: Biological: Peginterferon Alfa-2a; Drug: Ribavirin; Drug: Telaprevir

INTERVENTIONS:
Biological: Peginterferon Lambda-1a
  Other Names: BMS-914143
  Arms: Peginterferon Lambda-1a + Ribavirin + Daclatasvir
Biological: Peginterferon Alfa-2a
  Other Names: Pegasys®
  Arms: Peginterferon Alfa-2a + Ribavirin + Telaprevir
Drug: Ribavirin
  Other Names: Copegus®
Drug: Daclatasvir
  Other Names: BMS-790052
  Arms: Peginterferon Lambda-1a + Ribavirin + Daclatasvir
Drug: Telaprevir
  Other Names: Incivek®
  Arms: Peginterferon Alfa-2a + Ribavirin + Telaprevir

SUMMARY:
The purpose of this study is to determine if treatment with Pegylated Interferon Lambda-1a, given in combination with Ribavirin and Daclatasvir for 24 weeks, is as safe and effective as the standard treatment with Pegylated Interferon Alfa-2a + Ribavirin + Telaprevir in subjects who are infected with Chronic Hepatitis C virus genotype 1b and have never received any prior anti-HCV treatment, or who have relapsed after an initial, successful treatment with Pegylated Interferon Alfa + Ribavirin

ELIGIBILITY:
Inclusion Criteria:

* Patients chronically infected with HCV Genotype-1b
* Naïve to prior treatment or documented evidence of relapse after completion of the prescribed duration of treatment (duration may be 24 or 48 weeks, to be determined based upon local guidelines)
* HCV RNA viral load ≥100,000 IU/mL at screening
* Patients with compensated cirrhosis are permitted

Exclusion Criteria:

* Infection with Hepatitis C virus (HCV) other than Genotype-1b
* Positive Hepatitis B surface antigen (HBsAg) or Human immunodeficiency virus (HIV)-1/HIV-2 antibody test at screening
* Evidence of chronic liver disease caused by diseases other than chronic HCV infection
* Current evidence of or history of variceal bleeding, hepatic encephalopathy, or ascites requiring diuretics or paracentesis or evidence of any of these findings on physical examination performed at screening
* Current or known history of cancer (except adequately treated in situ carcinoma of the cervix, or basal or squamous cell carcinoma of the skin) within 5 years prior to screening
* Current evidence or known history of decompensated cirrhosis based on radiologic criteria or biopsy results and clinical criteria
* Laboratory values:

  1. Hemoglobin <12.0 g/dL (males) or <11.0 g/dL (females)
  2. Platelets <90,000/mm3
  3. Total serum bilirubin ≥2 mg/dL (unless due to Gilbert's disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with Sustained Virologic Response at post-treatment follow-up Week 12 (SVR12) | Post treatment follow-up Week 12

SECONDARY OUTCOMES:
Proportion of subjects who achieve SVR12 in treatment-naive subjects | Post treatment follow-up Week 12
Proportion of subjects with rash related dermatologic events | Up to 12 weeks of treatment
Proportion of subjects who develop treatment emergent cytopenic abnormalities | Up to 48 Weeks
  Treatment emergent cytopenic abnormalities [anemia as defined by Hemoglobin (Hb) < 10 g/dL, and/or neutropenia as defined by absolute neutrophil count (ANC) < 750/mm3, and or thrombocytopenia as defined by platelets < 50,000/mm3]
Proportion of subjects with on-treatment interferon (IFN) associated flu like/musculoskeletal symptoms | Up to 48 Weeks
Proportion of subjects who achieve SVR24 [Hepatitis C virus (HCV) Ribonucleic acid (RNA) < Lower limit of quantitation (LLOQ)] at post-treatment follow-up Week 24 | Post treatment follow-up Week 24
  SVR24 = Sustained virologic response at post treatment follow-up Week 24
Proportion of subjects with adverse events (AEs), Serious adverse events (SAEs), dose reductions, and discontinuations due to AEs through end of follow-up | Maximum of 72 weeks
Proportion of subjects who achieve SVR12 with a 24-week treatment regimen | Post treatment follow-up Week 12
Proportion of subjects who achieve Extended rapid virologic response (eRVR) (HCV RNA < LLOQ target not detected at Weeks 4 and 12 of treatment) | Weeks 4 and 12 of treatment
Patient Health Questionnaire-9 (PHQ-9) score through end of follow-up | Maximum of 72 weeks
Proportion of subjects with treatment emergent laboratory abnormalities by toxicity grade through End of treatment (EOT) | Maximum of 72 weeks
Proportion of subjects with the following on-treatment interferon-associated neuropsychiatric symptoms through EOT | Maximum of 48 weeks
  Psychiatric symptoms (depression, irritability or insomnia)
Association of Single nucleotide polymorphism (SNPs) in Interleukin 28B (IL28B) (including rs12979860) or equilibrative nucleoside transporter 1 (ENT1) with clinical responses | Post-treatment follow-up Week 12
  For each SNP in each candidate gene, allele and genotype frequencies will be summarized by treatment regimen
Resistant variants associated with virologic failure through end of follow-up | Maximum of 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (65):
- United States (8):
  - Va Long Beach Healthcare System, Long Beach, California
  - Gastrointestinal Specialists Of Georgia Pc, Marietta, Georgia
  - Weill Cornell Medical College, New York, New York
  - Premier Medical Group Of The Hudson Valley, Pc, Poughkeepsie, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Texas Clinical Research Institute, Llc, Arlington, Texas
  - Medvamc, Houston, Texas
- Argentina (4):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Mar del Plata, Buenos Aires
  - Local Institution, Prov de Santa Fe, Santa Fe Province
- France (3):
  - Local Institution, Clichy
  - Local Institution, Grenoble
  - Local Institution, Villejuif
- Germany (5):
  - Local Institution, Berlin
  - Local Institution, Essen
  - Local Institution, Hamburg
  - Local Institution, Mannheim
  - Local Institution, München
- Israel (4):
  - Local Institution, Haifa
  - Local Institution, Tel Aviv
  - Local Institution, Tel Litwinsky
  - Local Institution, Zafed
- Italy (5):
  - Local Institution, Foggia
  - Local Institution, Messina
  - Local Institution, Modena
  - Local Institution, Pavia
  - Local Institution, Pisa
- Japan (17):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Kitakyushu, Fukuoka
  - Local Institution, Kitakyushu-shi, Fukuoka
  - Local Institution, Gifu, Gifu
  - Local Institution, Hiroshima, Hiroshima
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Kobe, Hyōgo
  - Local Institution, Higashiibaraki-gun, Ibaraki
  - Local Institution, Kawasaki-shi, Kanagawa
  - Local Institution, Yokohama, Kanagawa
  - Local Institution, Kumamoto, Kumamoto
  - Local Institution, Kyoto, Kyoto
  - Local Institution, Saga, Saga-ken
  - Local Institution, Minato-ku, Tokyo
  - Local Institution, Musashino-shi, Tokyo
  - Local Institution, Sumida-ku, Tokyo
  - Local Institution, Tanabe-shi, Wakayama
- Poland (4):
  - Local Institution, Bialystok
  - Local Institution, Lodz
  - Local Institution, Mysłowice
  - Local Institution, Wroclaw
- Russia (3):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Stavropol
- South Korea (2):
  - Local Institution, Busan
  - Local Institution, Seoul
- Spain (4):
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Santander
  - Local Institution, Zaragoza
- Taiwan (5):
  - Local Institution, Kaohsiung, Taiwan
  - Local Institution, Taichung
  - Local Institution, Tainan
  - Local Institution, Taipei
  - Local Institution, Taoyuan District
- Local Institution, London, Greater London, United Kingdom

REFERENCES:
- [Derived] Flisiak R, Kawazoe S, Znoyko O, Assy N, Gadano A, Kao JH, Lee KS, Zwirtes R, Portsmouth S, Dong Y, Xu D, Kumada H, Srinivasan S. Peginterferon Lambda-1a/Ribavirin with Daclatasvir or Peginterferon Alfa-2a/Ribavirin with Telaprevir for Chronic Hepatitis C Genotype 1b. J Interferon Cytokine Res. 2016 Nov;36(11):635-643. doi: 10.1089/jir.2015.0173. Epub 2016 Jun 21. PMID 27327078
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx